CLINICAL TRIAL: NCT04279652
Title: The Effects of Combined Exercise Program in Children Attention Deficit Hyperactivity Disorder
Brief Title: Exercise in Children Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Arzu Demircioğlu, PT, MSc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19032
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: ADHD; Exercise
Keywords: ADHD; Exercise; motor proficiency
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised exercise group (Experimental): The treatment program was determined as 3 sessions per week for 8 weeks and 60 minutes per session. The treatment program consists of 5 min warm-up exercises, 20 min aerobic exercise, 20 min balance-coordination exercises, 10 min strengthening exercises and 5 min cooling exercises.
  Interventions: Other: Combined exercise
- Home exercise group (Active Comparator): The exercise program, which is prepared for the individual, will be applied to the home exercise group with 60 minutes of 3 times a week.
  Interventions: Other: Combined exercise
- Control group (No Intervention): Children will not be included in any treatment program. The assessments will be done again 8 weeks later.

INTERVENTIONS:
Other: Combined exercise — Combined exercise program consists of 5 min warm-up exercises, 20 min aerobic exercise, 20 min balance-coordination exercises, 10 min strengthening exercises and 5 min cooling exercises.
  Arms: Home exercise group; Supervised exercise group

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a heterogeneous neurodevelopmental disorder characterized by carelessness, hyperactivity and impulsivity, in which genetic, social and physical factors play an important role. Few studies have revealed the physical activity levels and importance of children with ADHD, but there is no consensus on the components of the physical activity program such as intensity, frequency, and severity. The aim of the present study is to investigate the effect of combined exercise training on motor proficiency, physical fitness and cognitive status in children with ADHD.

DETAILED DESCRIPTION:
The aim of present study is to investigate the effect of combined exercise training on motor proficiency, physical fitness and cognitive status in children with ADHD. Children will be randomly divided into 3 groups, for 8 weeks the first group will undergo a combined exercise training under the supervision of a physiotherapist, while the second group will receive a home exercise program. children included in the third group will form the control group.

The following assessments will be applied at the beginning and end of treatment.

1. Revised Conners Parent Rating Scale Short Turkish Form
2. Powers and Challenges Survey
3. Edinburgh Hand Preference Survey
4. Two-minute walking test
5. Ten meter walking test
6. Munich Fitness Test
7. Bruininks-Oseretsky Motor Proficiency Test-2
8. Muscle strength evaluation
9. Dynamic Occupational Therapy Cognitive Assessment
10. Open-ended questions

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with ADHD according to DSM-V (The Diagnostic and Statistical Manual of Mental Disorders-V) diagnostic criteria,
* Being between the ages of 7-12,
* Right hand being dominant according to Edinburgh Hand Preference Questionnaire,
* After the purpose of the study and the procedures to be explained, both the child and his family agree to participate in the study,
* An appropriate drug treatment program has been organized by the psychiatrist,
* The absence of a contraindicated condition to exercise in physical and medical examination.

Exclusion Criteria:

* A major psychiatric and / or neurodevelopmental problem accompanying,
* A history of head injury or chronic neurological disease,
* Having additional medical diseases that require medication,
* Any changes made in the psychiatric drug treatment by the attending physician for the last 1 month,
* Have participated in a regular exercise program or sporting activity for the past 6 months.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Motor Proficiency | 45 minutes
  Motor proficiency will be evaluated The Bruininks-Oseretsky Test of Motor Proficiency Second Edition (BOT™-2). t contains subtests and challenging game-like tasks and is very easy to administer. the score of this test ranges from 0 to 322. Higher score indicates better motor proficiency
Cognitive assessment | 90 minutes
  Dynamic Occupational Therapy Cognitive Assessment (DOTCA-Ch) battery for children allows to evaluate cognitive skills in 5 main topics: orientation, spatial perception, praxis, visual-motor organization and thinking processes.
Physical Fitness | 15 minutes
  Munich Fitness Test

SECONDARY OUTCOMES:
Behavior Disorders | 5 minutes
  Conners Parent Rating Scale consists of 27 items in total. In this scale, questions are answered on a 4-point Likert scale. "Never", "rarely", "often" and "always" options are; It is scored as "0", "1", "2" and "3". High scores from the scale show the intensity of symptoms specific to destructive disorders
Behaviour characteristics | 5 minutes
  Strength and Difficulties Questionnaire - (SDQ) "contains 25 questions, some of which question positive and some negative behavior characteristics. Each sub-title can be evaluated within itself and a separate score can be obtained for each, as well as the sum of the first four titles and the" Total Strength Score ".
Hand dominance | 5 minutes
  Edinburgh Hand Preference Questionnaire was developed to determine the hand preferences of the persons.The sum of the right and left hand scores gives "Cumulative Total (TC)" and subtracting the left hand score from the right hand score gives "Difference score (F)". The result score is obtained by dividing the difference score by the cumulative total score and multiplying it by the face. Result score; It can be interpreted that if the person is less than 40, the person is left dominant, and between -40 and 40, each bilateral dominant, and if greater than 40, the person is right dominant.
gait endurance | 4 minutes
  2-minute walking test will be used to determine walking endurance. In this test, a distance of 50 feet (15.2 meters) in length is determined first. The evaluator marks each 10 foot long distance with markers, leaving a cone at the beginning and end of the total distance.
muscle strength | 10 minutes
  Isometric muscle strength will be evaluated by hand dynamometer. Care is taken to repeat 3 times at short intervals during measurements. The highest value will be used for analysis. 4 muscle groups, including shoulder abductors, grip strength, hip flexors and ankle dorsi flexors, will be evaluated bilaterally.
10 meter walking test | 2 minutes
  Walking speed
Open ended questions | 15 minutes
  these questions for social cooperation and behaviour

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No